CLINICAL TRIAL: NCT04528693
Title: The Effect of 12-week Circuit Training (Combination of Strength and Endurance Exercises) on Insulin Sensitivity and Vascular Endothelial Function in Women With Insulin Resistance
Brief Title: The Effect of 12-week Circuit Training on Insulin Sensitivity and Endothelial Function in Women With Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Marzena Ratajczak, assistant professor, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PoznanUPhyEd no. 4
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Insulin Resistance
Keywords: circuit training; combined training; endothelial function; insulin sensitivity; lipid metabolism; inflammation; myokines; plantar stifness; back pain
MeSH Terms: conditions — Insulin Resistance; Inflammation; Back Pain | interventions — Circuit-Based Exercise

STUDY DESIGN:
Intervention Model Description: The study is designed as a prospective randomized clinical trial where subjects are randomally allocated to intervention group (study) or non-intervention group (control).
Who Masked: Care Provider
Masking Description: The qualifying physician does not know which of the examined persons will be allocated in the intervention or in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 40 women with insulin resistance aged 25-45, BMI 18,5-29,9 will perform, for a period of 3 months, 3 times a week, strength training, interspersed with bouts of endurance exercise carried out on circuit machines integrated with the Milon computer software.
  Interventions: Behavioral: Circuit training (combination of strength and endurance exercises)
- Control (No Intervention): 40 women with insulin resistance aged 25-45, BMI 18,5-29,9 will be asked to maintain their current level of physical activity and their diet for a period of 3 months.

INTERVENTIONS:
Behavioral: Circuit training (combination of strength and endurance exercises) — The intervention will last 3 months, exercises will take place 3 times a week and will consist of strength exercises, interspersed with bouts of endurance exercise carried out on circuit machines integrated with the Milon computer software for a total of 30 minutes per session.
  Other Names: Circuit training on machines integrated with the Milon computer software
  Arms: Intervention

SUMMARY:
During the last 10 years many studies concerning the impact of physical training on whole-body insulin sensitivity have been published, but there is a lack of an extended investigation on the potential clinical benefits of novel circuit training-based on strength and endurance exercises-relating to the optimization of insulin sensitivity and vascular endothelial function. It is of interest to precisely determine the physiological and biochemical effects of circuit training. An important aspect of the planned research will be the analysis of the effects of physical training on the released during muscle contraction myokines capable of modulating various metabolic processes. We hypothesized that in studied participants 12 weeks of the novel form of training would result in improving insulin sensitivity and vascular endothelial function mainly via myokines released by contracting skeletal muscles.

The following questions will be asked: (1) whether the 12-week circuit training (combined strength and endurance exercises) performed by women with insulin resistance, improves insulin sensitivity, carbohydrate and lipid metabolism and promotes the efficiency of endothelial defense mechanisms? (2) whether the 12-week circuit training (combined of strength and endurance exercises) changes the concentrations of transcription factors regulating lipid and carbohydrate metabolism or the synthesis and/or secretion of myokines and adipokines in women with insulin resistance? (3) whether the 12-week strength training, interspersed with bouts of endurance exercise has a positive effect on cytokine profile? (4) whether there is a relationship between changes in body composition, HOMA-IR, and the level of myokines caused by physical training? (5) whether the 12-week circuit training reduces low back pain symptoms, plantar stifness and improve functioning of the patient in everyday life? A group of 80 women, aged 25 to 45 years, with diagnosed insulin resistance will participate in the planned study. Participants will be enrolled in the research program based on medical qualification. Before the intervention all women will have venous blood collected to determine fasting glucose, hemoglobin glycosylated (HbA1C) and insulin levels and insulin resistance by the homeostasis model assessment of insulin resistance (HOMA-IR) will be calculated. The inclusion criteria will be as follows: (1) women, age: 25-45 years, menstruating, (2) BMI 18,5-29,9 kg/m2, (3) insulin resistance based on HOMA-IR (cut-off point 2.5), (4) HbA1C ≤ 6.5%, (5) not contraindicated to physical activity. Participants meeting the inclusion criteria will be randomly divided into two groups. The first group of women will undergo circuit training, consisting of exercises performed on 7 machines arranged in a circuit. Thanks to the use of adequate software the machines will automatically adjust their parameters, such as seat height or resistance to the exercising person, and the training progress will be individually monitored. The planned training will last for 3 months, during which the patients will exercise 3 times a week for 30 minutes (2 circuits will be done during each session). The planned duration of the training session will be controlled (one minute for strength exercises, four minutes for endurance exercises and a 30-second break between each exercise). In the training group, one-repetition maximum exercise test (1RM) will be performed to determine the appropriate training load and later after the program to verify the increase in muscle strength. The range of maximum heart rate (HRmax) will also be determined in all exercising women. The second group of women, who will be asked to maintain their current level of physical activity and their diet for a period of 3 months will serve as a control group. Before and after the training program in all participants of the study pulse wave velocity, anthropometric parameters and body composition will be assessed. Concurrently venous blood will be taken to determine biochemical indicators related to carbohydrate and lipid metabolism, insulin resistance, vascular endothelium function, inflammation and adipocytokines and myokines. In both groups of women, the questioners concerning dietary intake and the level of daily physical activity will be administered.

Results will be subjected to analysis involving descriptive, and advanced statistic method among them analysis of correlations, regression, variance and cluster analysis. All calculations and statistics will be performed using TIBCO Statistica 13.3 software (TIBCO).

DETAILED DESCRIPTION:
The training program will be performed on 7 machinesin a circuit. The devices will be controlled by a pre-programmed chip card, so that they will automatically adjust their parameters, such as seat height or resistance to the patient, and it will be possible to monitor the training progress of exercising women and their presence during training. Only two people will be allowed in the room during the training. The planned duration of the exercises will be controlled (one minute for strength exercises, four minutes for endurance exercisesand a 30-second break between each exercise) and for each trainee the load will be dosed using the electronic resistance motor system. Exercises in the training program are planned in such a way that the different muscle groups of women exercising are loaded alternately, which will ensure comprehensive training of the whole body. The range of movement, exercise duration and breaks will be controlled automatically by the system and the software of the devices and will not require additional training attention.

In the training group, one-repetition maximum exercise test (1RM) will be performed to determine the appropriate training load and later after the program to verify the increase in muscle strength.

The HR max range will be determined for exercising women by the indirect method using the formula: training HR = 220 -subject age.

The characteristics of exercises in the circuit:

1. The training circuit starts with an exercise on a cycloergometer -"bike", which lasts 4 minutes.
2. The second exercise -"abdominal crunch", shapes the strength of the abdominal muscles and together with exercise number six, it not only improves muscle strength parameters, but also shapes balance and maintains the correct position of the body.
3. The third exercisein a circuit-"leg curl", shapes the muscular strength of the back of the thigh (biceps femoris muscleand muscles adjacent to it).
4. The fourth exercise -"lat pulldown", trains the strength of the latissimus dorsi muscle, shoulder girdle muscles and upper chest. In addition to improving the strength and function of the muscles mentioned above, the exercise also perfectly stimulates the auxiliary respiratory muscles.
5. Fifth exercise -"crosswalker".This exercise trainsmost of the body's muscles, itlasts 4 minutes and, like training on a cycloergometer, primarily shapes thephysical capacity.
6. The sixth exercise -"back extension"trains the strength of the abdominal muscles, erector spinae and other muscles of a back.
7. The seventh exercise -"legabductor", the last in the series, is an exercise that shapes the gluteal muscles, as well as hip adductor and abductor muscles. This exercise fulfills the function of shaping strength and securing the hip joint, by training the muscle parts less frequently used in everyday life, the more difficult to be kept fit as the years go by and the level of physical activity decreases.

ELIGIBILITY:
Inclusion Criteria:

* women,
* age: 25-45years,
* menstruating,
* BMI 18,5-29,9 kg/m2,
* insulin resistance based on HOMA -IR (cut-off point 2.5),
* not contraindicated to physical activity.

Exclusion Criteria:

* type 1 and 2 diabetes,
* poorly controlled hypertension (mean SBP >140mmHg and/or mean DBP >90mmHg) over the last month and/or need to modify the pharmacological treatment,
* obesity: BMI > 30 kg/m2,
* lipid disorders requiring implementation of pharmacological treatment in the last 3 months before or during observation,
* a positive history of ischemic heart disease, carotid atherosclerosis and / or lower limb atherosclerosis,
* clinically significant arrhythmias or conduction disorders,
* chronickidney disease,
* clinically significant liver dysfunction,
* acute or chronic, clinically manifest inflammatory process,
* an acute infection in the last month,
* cancer,
* taking dietary supplements within a month before inclusion and during observation,
* taking medication that could interfere with the results of the tests,
* other conditions that may pose any risk to the patient during the observation.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Homeostasis model assessment of insulin resistance (HOMA-IR) | pre-intervention
Homeostasis model assessment of insulin resistance (HOMA-IR) | 48 hours after the intervention
HbA1C [mmol/mol] | pre-intervention
  ELISA
HbA1C [mmol/mol] | 48 hours after the intervention
  ELISA
Insuline [mU/ml] | pre-intervention
  Radioimmunoassay
Insuline [mU/ml] | 48 hours after the intervention
  Radioimmunoassay
Systolic and diastolic blood pressure [mmHg] | pre-intervention
Systolic and diastolic blood pressure [mmHg] | 48 hours after the intervention
Pulse wave velocity (PWV) [m/s] | pre-intervention
  PWV will be performed using the SphygmoCor Px (Atcor Medical Blood Pressure Analysis System, Sydney, Australia.
Pulse wave velocity (PWV) [m/s] | 48 hours after the intervention
  PWV will be performed using the SphygmoCor Px (Atcor Medical Blood Pressure Analysis System, Sydney, Australia.
Glucose, Total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) and triglycerides (TG) [mmol/l] | pre-intervention
  Dimension Flex Reagent Cartridge
Glucose, Total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) and triglycerides (TG) [mmol/l] | 48 hours after the intervention
  Dimension Flex Reagent Cartridge
Irisin, Visfatin, Retinol-binding protein 4 (RBP-4) [pg/ml] | pre-intervention
  ELISA
Irisin, Visfatin, Retinol-binding protein 4 (RBP-4) [pg/ml] | 48 hours after the intervention
  ELISA
Apelin [ng/ml] | pre-intervention
  ELISA
Apelin [ng/ml] | 48 hours after the intervention
  ELISA
C Reactive Protein (hsCRP) [mg/l] | pre-intervention
  ELISA
C Reactive Protein (hsCRP) [mg/l] | 48 hours after the intervention
  ELISA
Interleukin-6 (IL-6), Interleukin-10 (IL-10) [pg/ml] | pre-intervention
  ELISA
Interleukin-6 (IL-6), Interleukin-10 (IL-10) [pg/ml] | 48 hours after the intervention
  ELISA
Endothelial nitric oxide synthase (eNOS) [ng/ml] | pre-intervention
  ELISA
Endothelial nitric oxide synthase (eNOS) [ng/ml] | 48 hours after the intervention
  ELISA
Muscle strength [kg] | pre-intervention
  Test 1RM will be performed for following groups of muscles: abdominal muscles; back of the thigh (biceps femoris muscle and muscles adjacent to it); latissimus dorsi muscle, shoulder girdle muscles and upper chest; erector spinae and other muscles of a back; gluteal muscles, hip adductor and abductor muscles.
Muscle strength [kg] | 48 hours after the intervention
  Test 1RM will be performed for following groups of muscles: abdominal muscles; back of the thigh (biceps femoris muscle and muscles adjacent to it); latissimus dorsi muscle, shoulder girdle muscles and upper chest; erector spinae and other muscles of a back; gluteal muscles, hip adductor and abductor muscles.

SECONDARY OUTCOMES:
Plantar stiffness [N/m] | pre-intervention
  Biomechanical properties will be assessed with myotonometer device.
Plantar stiffness [N/m] | 48 hours after the intervention
  Biomechanical properties will be assessed with myotonometer device.
State of tension of erector spinae muscles [Hz] | pre-intervention
  Natural oscillation frequency [Hz], characterizing Tone or Tension will be assessed with myotonometer device.
State of tension of erector spinae muscles [Hz] | 48 hours after the intervention
  Natural oscillation frequency [Hz], characterizing Tone or Tension will be assessed with myotonometer device.
Low back pain intensity: questionnaire | pre-intervention
  Visual analogue scale (VAS) pain intensity questionare (reporting a score on a 10-point scale, the minimum (0) means no pain and the maximum (10) means a worst pain imaginable
Low back pain intensity: questionnaire | 48 hours after the intervention
  Visual analogue scale (VAS) pain intensity questionare (reporting a score on a 10-point scale, the minimum (0) means no pain and the maximum (10) means a worst pain imaginable
Disability caused by pain in the spine | pre-intervention
  Oswestry questionnaire. When completing the questionnaire, the subject answers questions concerning: pain intensity, independence, lifting objects, walking, sitting, standing, sleeping, social life, sexual activity and traveling. The answers to the questions help to classify how limited the functioning of the patient is while performing certain activities. Responses are graded from 0 to 5. The overall score is given on a 0-50 point scale, where the higher the score, the greater the disability.
Disability caused by pain in the spine | 48 hours after the intervention
  Oswestry questionnaire. When completing the questionnaire, the subject answers questions concerning: pain intensity, independence, lifting objects, walking, sitting, standing, sleeping, social life, sexual activity and traveling. The answers to the questions help to classify how limited the functioning of the patient is while performing certain activities. Responses are graded from 0 to 5. The overall score is given on a 0-50 point scale, where the higher the score, the greater the disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Srikanthan P, Karlamangla AS. Relative muscle mass is inversely associated with insulin resistance and prediabetes. Findings from the third National Health and Nutrition Examination Survey. J Clin Endocrinol Metab. 2011 Sep;96(9):2898-903. doi: 10.1210/jc.2011-0435. Epub 2011 Jul 21. PMID 21778224
- [Background] Bird SR, Hawley JA. Update on the effects of physical activity on insulin sensitivity in humans. BMJ Open Sport Exerc Med. 2017 Mar 1;2(1):e000143. doi: 10.1136/bmjsem-2016-000143. eCollection 2016. PMID 28879026
- [Background] Lambers S, Van Laethem C, Van Acker K, Calders P. Influence of combined exercise training on indices of obesity, diabetes and cardiovascular risk in type 2 diabetes patients. Clin Rehabil. 2008 Jun;22(6):483-92. doi: 10.1177/0269215508084582. PMID 18511528
- [Background] Oh KJ, Lee DS, Kim WK, Han BS, Lee SC, Bae KH. Metabolic Adaptation in Obesity and Type II Diabetes: Myokines, Adipokines and Hepatokines. Int J Mol Sci. 2016 Dec 22;18(1):8. doi: 10.3390/ijms18010008. PMID 28025491
- [Background] Ormazabal V, Nair S, Elfeky O, Aguayo C, Salomon C, Zuniga FA. Association between insulin resistance and the development of cardiovascular disease. Cardiovasc Diabetol. 2018 Aug 31;17(1):122. doi: 10.1186/s12933-018-0762-4. PMID 30170598
- [Derived] Karolkiewicz J, Krzywicka M, Szulinska M, Musialik K, Musialowska D, Zielinski J, Bilska A, Ratajczak M. Effects of a Circuit Training Program on Myokine Levels in Insulin-Resistant Women: A Randomised Controlled Trial. J Diabetes Res. 2024 Nov 28;2024:6624919. doi: 10.1155/jdr/6624919. eCollection 2024. PMID 39640300
- [Derived] Ratajczak M, Krzywicka M, Szulinska M, Musialowska D, Kusy K, Karolkiewicz J. Effects of 12-Week Combined Strength and Endurance Circuit Training Program on Insulin Sensitivity and Retinol-Binding Protein 4 in Women with Insulin-Resistance and Overweight or Mild Obesity: A Randomized Controlled Trial. Diabetes Metab Syndr Obes. 2024 Jan 6;17:93-106. doi: 10.2147/DMSO.S432954. eCollection 2024. PMID 38204866